CLINICAL TRIAL: NCT05487183
Title: Test Retest Reliability of Offset Analgesia and Onset Hyperalgesia Paradigm
Brief Title: Test Retest Reliability of OA and OH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Benedict Alter, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY22010185
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Analgesia; Pain Catastrophizing; Pain
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): QST devices and computer tasks are used to measure OA, OH, pain intensity, and other outcomes
  Interventions: Behavioral: Medoc cutaneous probe; Behavioral: Quantitative sensory testing; Behavioral: Computer tasks

INTERVENTIONS:
Behavioral: Medoc cutaneous probe — A computer-controlled probe delivers temperatures to the skin to measure pain, OA, and OH
Behavioral: Quantitative sensory testing — Standard methods involving pinprick, pressure, heat, and cold applied to the skin are used to measure sensation and pain
Behavioral: Computer tasks — QST and computer tasks are used to measure changes in pain intensity

SUMMARY:
The goal of this study is to measure the test retest reliability of offset analgesia (OA) and onset hyperalgesia (OH) across multiple study visits. OA and OH are quantitative sensory tests (QST) thought to measure how the brain modulates pain. This study will use a heat thermode to induce OA and OH in healthy, pain-free volunteers across 3 study visits. Additional QST measures and survey data relevant to pain modulation will be collected. This study lays the foundation required to use OA and OH as tools to measure pain modulation in clinical trials. Following their validation, we anticipate that OA and OH will serve as predictive and therapeutic biomarkers, which will aid both in the development of novel analgesics and in treatment selection leading to the personalization of pain management.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with no chronic pain issues who can understand the study procedures

Exclusion Criteria:

* History of chronic pain
* Current significant pain disorder
* Active ongoing pain every day that is acute or chronic in duration
* Recent history of migraine (1 attack in last 24 months)
* Lifetime history mood disorders (anxiety, depression, bipolar) or psychotic disorders.
* Subjects taking psychotropics (e.g. benzodiazepines, antidepressants), or medications known to affect the autonomic nervous system (e.g. beta-receptor agonists or antagonists) will be excluded.
* Cognitive impairment affecting the ability to provide informed consent, understand directions, and participate in study procedures
* Uncontrolled or unstable medical disorder preventing participation in study procedures
* Pregnancy
* Tattoos on forearm
* History of brain surgery
* Nonambulatory status
* Heart problems such as an irregular heart beat or coronary artery disease
* Neurological problems such as seizure, fainting spells, recurrent severe headache, stroke, transient ischemic attack
* High blood pressure
* Severe liver disease
* Severe gastrointestinal disease
* Chronic severe infectious disease (e.g. HIV/AIDS)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Offset analgesia and onset hyperalgesia | baseline
  Pain intensity difference during heat stimuli measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable) at baseline
Test retest reliability of offset analgesia and onset hyperalgesia | 1 week post baseline
  Pain intensity difference during heat stimuli measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable) at 1 week after baseline
Test retest reliability of offset analgesia and onset hyperalgesia | 4 weeks post baseline
  Pain intensity difference during heat stimuli measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable) at 4 weeks after baseline
Differences in brain region activation- QST (quantitative sensory tests) | baseline
  Difference in brain region activation (as measured by oxygenated hemoglobin, HbO) between central nervous system inhibition and control stimuli during QST procedures.
Test retest reliability in brain region activation- QST (quantitative sensory tests) | 1 week post baseline
  Difference in brain region activation (as measured by oxygenated hemoglobin, HbO) between central nervous system inhibition and control stimuli during QST procedures at 1 week after baseline
Test retest reliability in brain region activation- QST (quantitative sensory tests) | 4 weeks post baseline
  Difference in brain region activation (as measured by oxygenated hemoglobin, HbO) between central nervous system inhibition and control stimuli during QST procedures at 4 weeks after baseline

SECONDARY OUTCOMES:
Differences in resting fNIRS signaling | baseline
  Differences in fNIRS resting state connectivity as measured by brain region activation
Questionnaire score- State Trait Anxiety Inventory (STAI) Y1-2 | baseline
  Standardized survey score of state trait anxiety inventory Y1 and Y2 assessing anxiety before QST procedures on visit 1 only.
  State Anxiety Score ranges from 20-80. Trait Anxiety Score ranges from 20-80. Higher scores indicate worse anxiety state and trait symptoms.
Questionnaire score- Pain Catastrophizing Scale (PCS) | baseline
  Standardized survey score assessing pain perception before QST procedures at visit 1 only. Rumination subscale score ranges from 0-16. Magnification subscale score ranges 0-12. Helplessness subscale score ranges from 0-24. Total score can be calculated by summing subscales. Total score ranges from 0-52, with higher scores indicating more pain catastrophizing.
Questionnaire score- STAI Y1 post testing | baseline
  Standardized survey score of state trait anxiety inventory Y1 assessing anxiety immediately after QST procedures measured at all 3 visits. Higher scores indicate worse anxiety state.
Questionnaire score- STAI Y1 post testing | 1 week after baseline
  Standardized survey score of state trait anxiety inventory Y1 assessing anxiety immediately after QST procedures measured at all 3 visits. Higher scores indicate worse anxiety state.
Questionnaire score- STAI Y1 post testing | 4 weeks after baseline
  Standardized survey score of state trait anxiety inventory Y1 assessing anxiety immediately after QST procedures measured at all 3 visits. Higher scores indicate worse anxiety state.
Questionnaire score- Situational Pain Catastrophizing Scale post testing | baseline
  Standardized survey score assessing pain perception immediately after QST procedures are completed at each visit.
  Scores range from 0-24, with higher scores representing more pain catastrophizing.
Questionnaire score- Situational Pain Catastrophizing Scale post testing | 1 week after baseline
  Standardized survey score assessing pain perception immediately after QST procedures are completed at each visit.
  Scores range from 0-24, with higher scores representing more pain catastrophizing.
Questionnaire score- Situational Pain Catastrophizing Scale post testing | 4 weeks after baseline
  Standardized survey score assessing pain perception immediately after QST procedures are completed at each visit.
  Scores range from 0-24, with higher scores representing more pain catastrophizing.
Questionnaire score- Beck Depression Inventory-II (BDI-II) | baseline
  Standardized survey assessing depression at the start of visit 1. Scores range from 0-63. Total score of 0-13 is considered minimal range of depression, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
Questionnaire score- Generalized Anxiety Disorder 2-item (GAD-2) | baseline
  Standardized survey score of GAD-2 assessing anxiety at the start of visit 1. Scores range from 0-6. Higher scores indicate higher likelihood of having GAD.
Questionnaire score- Multidimensional Assessment of Interoceptive Awareness (MAIA) Version 2 | baseline
  Standardized survey score of MAIA-2 assessing mindfulness at the start of visit 1. Total scores range from 0-160 with 8 subscales. Higher scores indicate higher levels of mindfulness.
Questionnaire score- Multidimensional Assessment of Interoceptive Awareness (MAIA) Version 2 post testing | baseline
  Standardized survey score of MAIA-2 assessing mindfulness after QST measured at all 3 visits. Total scores range from 0-160 with 8 subscales. Higher scores indicate higher levels of mindfulness.
Questionnaire score- Multidimensional Assessment of Interoceptive Awareness (MAIA) Version 2 post testing | 1 week after baseline
  Standardized survey score of MAIA-2 assessing mindfulness after QST measured at all 3 visits. Total scores range from 0-160 with 8 subscales. Higher scores indicate higher levels of mindfulness.
Questionnaire score- Multidimensional Assessment of Interoceptive Awareness (MAIA) Version 2 post testing | 4 weeks after baseline
  Standardized survey score of MAIA-2 assessing mindfulness after QST measured at all 3 visits. Total scores range from 0-160 with 8 subscales. Higher scores indicate higher levels of mindfulness.
Pain intensity | baseline
  Changes in pain intensity during quantitative sensory tests and computer tasks measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable)
Pain intensity | 1 week after baseline
  Changes in pain intensity during quantitative sensory tests and computer tasks measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable)
Pain intensity | 4 weeks after baseline
  Changes in pain intensity during quantitative sensory tests and computer tasks measured on a 0-100 sliding scale (0 is no pain, 100 is the most intense pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Alter, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Pain Medicine at Centre Commons, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available, including data dictionaries, after publication per journal and funding protocols. The statistical analysis plan and analytic code will also be available per the same protocols.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after publication per journal and funding entity protocols.
Access Criteria: Data will be made available by reasonable request and/or per journal and funding entity protocols.